CLINICAL TRIAL: NCT01288144
Title: Clinical Decision Support for Women With a History of Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ellen W. Seely, M.D., Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2007p000842
Record Dates: First submitted 2010-08-25; First posted 2011-02-02 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Screening; Gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Quality improvement initiative using computerized decision support
  Interventions: Other: Quality improvement initiative
- Usual care (No Intervention): In control clinics, women will continue to receive usual care.

INTERVENTIONS:
Other: Quality improvement initiative — In intervention clinics, the LMR will use the existing reminder function to alert providers that a patient has a probable history of gestational diabetes. The provider will then have the opportunity to clarify the subject's history and order appropriate screening testing. Providers will also have access to online reference material regarding GDM follow-up screening and lifestyle interventions.
  Other Names: Quality improvement initiative using computerized decision support
  Arms: Intervention

SUMMARY:
The investigators hypothesize that computer-assisted decision support will increase the percentage of women with a history of gestational diabetes who receive appropriate follow-up screening.

Specific Aim 1: Develop an algorithm to identify cases of gestational diabetes among patients in the Partners Health Care system using administrative and laboratory data.

Specific Aim 2: Assess primary care provider knowledge, attitudes, beliefs, and barriers to compliance regarding screening guidelines for women with a history of gestational diabetes.

Specific Aim 3: Test whether a computer-assisted decision support tool to identify patients with a GDM history and prompt screening will increase compliance with guidelines. The investigators hypothesize that decision support will significantly increase in the percentage of women screened.

DETAILED DESCRIPTION:
Approximately 5 percent of women are diagnosed with gestational diabetes (GDM) during pregnancy. These women face an increased risk of progression to type 2 diabetes1 and may benefit from lifestyle interventions and screening to detect early disease. However, studies have shown that less than half of women are screened appropriately in the postpartum period. This performance gap may reflect both lack of communication between obstetric and primary care providers and lack of knowledge of appropriate screening guidelines. The investigators plan to assess a quality improvement initiative, using administrative and clinical data, to identify women with a history of GDM and implement decision support to enhance quality of care.

ELIGIBILITY:
Inclusion:

* Primary care clinic (gynecology, internal medicine, community health center)
* Use longitudinal medical record (LMR) program for documentation
* Previously participated in rct of decision support intervention

Exclusion:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2007-07; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Rate of screening | 1 year following implementation at all sites (Nov. 2011)
  The American Diabetes Association recommends that women with a history of GDM undergo glucose screening at 6 weeks post partum. Women with normal postpartum glucose testing should receive follow-up testing every three years, and those with impaired glucose tolerance should receive annual follow-up screening.
  Our study will evaluate a quality improvement intervention to increase the number of women who are appropriately identified and undergo screening.

REFERENCES:
- [Derived] Zera CA, Bates DW, Stuebe AM, Ecker JL, Seely EW. Diabetes Screening Reminder for Women With Prior Gestational Diabetes: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):109-14. doi: 10.1097/AOG.0000000000000883. PMID 26241263